CLINICAL TRIAL: NCT02797184
Title: Inorganic NItrate and EXercise Performance in Heart Failure (iNIX-HF): Dose Response
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016_11111
Record Dates: First submitted 2016-05-25; First posted 2016-06-13 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — potassium nitrate

STUDY DESIGN:
Intervention Model Description: Subjects will receive one drug dose on the first dose visit and the second drug dose on the second dose visit. The order of the two drug doses (10 and 20 mmol KNO3) will be randomized, so that some subjects will receive the lower dose first and others will receive the higher dose first
Who Masked: Participant, Investigator
Masking Description: Both the participant and the investigator will be masked to which KNO3 dose is administered at each visit. However, it is known at the outset that each patient will receive 10 mmol KNO3 during one visit and 20 mmol KNO3 at another visit, with the order randomly assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10mmol KNO3 (Experimental): Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (10 or 20 mmol KNO3) in 2 gelatin capsules during dose visit 1 and the other dose (10 or 20 mmol KNO3) during dose visit 2. The dose order will be randomized.
  Interventions: Drug: KNO3, potassium nitrate
- 20mmol KNO3 (Experimental): Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (10 or 20 mmol KNO3) in 2 gelatin capsules during dose visit 1 and the other dose (10 or 20 mmol KNO3) during dose visit 2. The dose order will be randomized.
  Interventions: Drug: KNO3, potassium nitrate

INTERVENTIONS:
Drug: KNO3, potassium nitrate — Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
  Other Names: saltpeter

SUMMARY:
The purpose of this study is to do the work that is necessary and sufficient for setting up an appropriate multi-center, randomized clinical trial (RCT) of a new therapy for heart failure: inorganic nitrate. The investigators will first determine the effects and palatability of ~12.8mmol KNO3 (an oral pill) as compared to the roughly equivalent amount of nitrate in 2 beetroot juice (BRJ) Sports Shots (by James White Drinks). Next, the investigators will determine the effects of inorganic nitrate (KNO3 in an oral pill format) on blood pressure, blood nitrate levels, breath nitric oxide (NO) levels, and exercise performance in a dose-response study. Third, the investigators will perform a small phase II chronic treatment study that will allow them to determine the best primary endpoint and the numbers of patients the investigators will need to study in the large, multi-center RCT to follow this project. In the small study and in the RCT to follow, the investigators will determine whether inorganic nitrate can improve aerobic exercise capacity, muscle power, and speed of muscle contraction, and lessen the effort of breathing during exercise.

DETAILED DESCRIPTION:
1. Subjects will be patients with Heart Failure (HF).
2. All subjects will be consented.
3. All subjects will give permission for the investigators to review their medical records.
4. After consenting to participate, subjects will be instructed to refrain from spitting or the use of an antibacterial mouthwash, antacids, proton pump inhibitors, or chewing gum during the morning of each clinic visit.
5. Subjects will have a physical examination.
6. Subjects will undergo transthoracic echocardiographic imaging at rest (unless they had this performed within the past 6 months).
7. Subjects will be asked to undergo a mouth swab for bacterial DNA analyses.
8. Subjects will be asked to answer questionnaires regarding their medical health (basic health questionnaire, Minnesota living with heart failure questionnaire, a combined fatigue questionnaire.
9. Dose visit 1: Subjects will receive 2 capsules containing either 10 or 20 mmol of potassium nitrate (KNO3).
10. Before and at 3 hourly time points after receiving the KNO3, subjects will undergo phlebotomy for plasma nitrite levels, will have their blood pressure measured, and will blow into a small machine to assess the amount of nitric oxide in their breath.
11. Exercise Test 1: Subjects will complete measurements of leg muscle power by doing knee extension exercises on a dynamometer (a device that measures voluntary muscle force production while controlling the speed of movement).
12. Exercise Test 2: Subjects complete a measurement of peak aerobic capacity (VO2peak) while walking on a treadmill and breathing into a mouthpiece. Blood pressure, heart rate and heart rhythm will be monitored during this test.
13. Subjects will undergo a 7 d washout period.
14. Dose visit 2: Subjects will receive 2 capsules containing either 10 or 20 mmol of KNO3 (whichever dose they did not receive at dose visit 1). They will repeat the same assessments listed above in 10, 11, and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: females and males
2. Age: at least 18 years and less than 75 years
3. Diagnosis of heart failure with reduced ejection fraction (NYHA II-IV)
4. Ejection fraction <45% as determined on an imaging study within 12 mo of enrollment
5. Stable medical therapy - defined by no addition or removal (or change of more than 100%) of the following: beta-adrenergic blockade, angiotensin converting enzyme (ACE) inhibitors, or angiotensin receptor blocker (ARB or aldosterone antagonists) for 30 days prior to enrolment

Exclusion Criteria:

1. "Vulnerable populations" as defined by the U.S. Department of Health and Human Services, such as prisoners and children
2. Pharmacologic, organic nitrate therapy within the last 3 months
3. Major orthopedic, psychiatric, neurological, or other conditions that would impair performance of the exercise tests in this study
4. Atrial fibrillation/flutter
5. Estimated glomerular filtration rate < 50 ml/min on most recent clinical laboratories
6. Systolic blood pressure < 95 mmHg or >180 mmHg at consent
7. Diastolic blood pressure <40 mmHg or >100 mmHg at consent
8. Previous adverse reaction to nitrates necessitating withdrawal of therapy
9. Treatment with phosphodiesterase inhibitors within the last 3 months (patient must also be willing to not take them for the duration of the trial).
10. Ejection fraction > 45%
11. Primary hypertrophic cardiomyopathy
12. Infiltrative cardiomyopathy (e.g., amyloid)
13. Active myocarditis
14. Complex congenital heart disease
15. Active collagen vascular disease
16. Active angina/ischemia from epicardial coronary disease
17. Percutaneous coronary intervention, new bi-ventricular pacing, or coronary artery bypass grafting within the past 3 months
18. More than mild mitral or aortic stenosis
19. Valvular heart disease with severe regurgitation of any valve.
20. Acute or chronic severe liver disease as evidenced by encephalopathy, international normalized ratio (INR) >1.7 without anticoagulation therapy, or variceal bleeding
21. Patients requiring exogenous oxygen at rest or for exercise
22. Terminal disease (other than heart failure) with expected survival < 1 y
23. Enrollment in another therapeutic trial during the period of the study
24. Pregnancy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine; Andrew R Coggan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
HIPPA-related data will not be available for publishing. Study results will be published in accordance with journal, institution, and HIPPA guidelines.

RESULTS

PARTICIPANT FLOW:
Groups:
- 10mmol KNO3, Then 20mmol KNO3: Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (10mmol KNO3) in 2 gelatin capsules during dose visit 1 and the otherv20 mmol KNO3 during dose visit 2.
  KNO3, potassium nitrate: Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
- 20mmol KNO3, Then 10mmol KNO3: Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (20 mmol KNO3) in 2 gelatin capsules during dose visit 1 and 10mmol KNO3 during dose visit 2.
  KNO3, potassium nitrate: Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
Period: Overall Study
Arm/Group | 10mmol KNO3, Then 20mmol KNO3 | 20mmol KNO3, Then 10mmol KNO3
Started | 21 | 21
Completed | 3 | 3
Not Completed | 18 | 18
Not completed — Study was put on hold due to COVID-19. Could not finish these subjects before funding ran out. | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (10 or 20 mmol KNO3) in 2 gelatin capsules during dose visit 1 and the other dose (10 or 20 mmol KNO3) during dose visit 2. The dose order will be randomized.
  KNO3, potassium nitrate: Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: VO2peak
Description: peak oxygen consumption during treadmill exercise
Time Frame: acute - 2.5 hours post dose
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | 10mmol KNO3 | 20mmol KNO3
Number analyzed (Participants) | 6 | 6
mL/kg/min | 17.7 (3.4) | 18.0 (4.1)

2. Secondary Outcome: Peak Muscle Power
Description: Participants completed measurements of leg muscle power by doing knee extension exercises on a dynamometer (a device that measures voluntary muscle force production while controlling the speed of movement).
Time Frame: acute - 2 hours post dose
Measure: Mean (Standard Deviation); unit: Watts/kg
Arm/Group | 10mmol KNO3 | 20mmol KNO3
Number analyzed (Participants) | 6 | 6
Watts/kg | 469.4 (188.8) | 497.9 (173.8)

3. Secondary Outcome: Blood Nitrite Levels
Description: concentrations of nitrite in the blood
Time Frame: time 0 (before receiving the KNO3 dose) and hourly after receiving KNO3 (1, 2, and 3 hours post-dose)
Measure: Mean (Standard Deviation); unit: micro M
Arm/Group | 10mmol KNO3 | 20mmol KNO3
Number analyzed (Participants) | 6 | 6
micro M
  0 hr | 0.489 (0.295) | 0.432 (0.258)
  1 hr post-ingestion KNO3 | 0.568 (0.244) | 0.591 (0.481)
  2 hr post-ingestion KNO3 | 0.658 (0.277) | 0.864 (0.916)
  3 hr post-ingestion KNO3 | 0.646 (0.261) | 0.769 (0.529)

4. Secondary Outcome: Breath Nitric Oxide (NO) Level
Description: Breath nitric oxide (NO) level will be taken via NIOX breath analyzer
Time Frame: time 0 (before receiving the KNO3 dose) and hourly after receiving KNO3 (1, 2, and 3 hours post-dose)
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | 10mmol KNO3 | 20mmol KNO3
Number analyzed (Participants) | 4 | 4
ppb
  0 hr | 26 (13) | 23 (9)
  1 hr | 28 (11) | 30 (14)
  2 hr | 28 (9) | 36 (21)
  3 hr | 32 (7) | 43 (16)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study period (about 6 weeks)
Groups:
- 10mmol KNO3: Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (10 mmol KNO3) in 2 gelatin capsules during dose visit 1 and the other dose (20 mmol KNO3) during dose visit 2. The dose order will be randomized.
  KNO3, potassium nitrate: Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
- 20mmol KNO3: Intervention: Subjects with heart failure will receive a single oral dose of potassium nitrate (20 mmol KNO3) in 2 gelatin capsules during dose visit 1 and the other dose (10 mmol KNO3) during dose visit 2. The dose order will be randomized.
  KNO3, potassium nitrate: Potassium nitrate (KNO3) will be given orally in 2 gelatin capsules, which will be compounded by the Barnes-Jewish Hospital Pharmacy. The doses are 10 mmol and 20 mmol KNO3.
Arm/Group | 10mmol KNO3 | 20mmol KNO3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT02797184/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02797184/ICF_001.pdf